CLINICAL TRIAL: NCT02147431
Title: A Randomised, Single-centre, Double-blind, Cross-over Trial Investigating the Effect of Semaglutide on Hypoglycaemic Counter-regulation Compared to Placebo in Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Effect of Semaglutide on Hypoglycaemic Counterregulation Compared to Placebo in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3684; 2013-002751-15 (EudraCT Number); U1111-1144-7019 (Other: WHO)
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — 2 periods of 12 weeks of once weekly dosing with multiple doses of semaglutide, for subcutaneous (s.c., under the skin) injection, escalated up to 1.0 mg semaglutide.
  Each treatment period will be followed by a hypoglycaemic clamp
  Arms: Semaglutide
Drug: placebo — 2 periods of 12 weeks of once weekly dosing, subcutaneous (s.c., under the skin) injection.
  Each treatment period will be followed by a hypoglycaemic clamp.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the effect of semaglutide on hypoglycaemic counter-regulation compared to placebo in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes and on stable treatment for a period of 90 days prior to screening with metformin as monotherapy. Stable is defined as unchanged dose
* Male or female, age between18-64 years (both inclusive) at the time of signing informed consent
* Body Mass Index (BMI) between 20.0-35.0 kg/m^2 (both inclusive)
* HbA1c (glycosylated haemoglobin) between 6.5-10.0% (both inclusive)

Exclusion Criteria:

* Treatment with any glucose lowering agent(s) other than metformin in a period of 90 days before screening. An exception is short-term treatment (less than or equal to 7 days in total) with insulin in connection with intercurrent illness
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Blood or plasma donation within the past month or more than 500 mL within the last 3 months prior to first semaglutide dosing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2015-05-20 (Actual)

PRIMARY OUTCOMES:
Change in mean glucagon concentration during hypoglycaemia (change from target level 5.5 mmol/L to nadir (target 2.5 mmol/L)) | After 12 weeks 2 days of treatment in each treatment period (Day 87 and Day 213)

SECONDARY OUTCOMES:
Change in mean glucagon concentration from target level 5.5 mmol/L to 3.5 mmoL/L and from ambient plasma glucose to target levels 5.5 mmol/L, 3.5 mmol/L and nadir | After 12 weeks 2 days of treatment in each treatment period (Day 87 and Day 213)
Change in mean concentrations of adrenaline, noradrenaline, cortisol and growth hormone from target level 5.5 mmol/L to 3.5 mmol/L and to nadir | After 12 weeks 2 days of treatment in each treatment period (Day 87 and Day 213)
Hypoglycaemic symptoms score | After 12 weeks 2 days of treatment in each treatment period (Day 87 and Day 213)
Time from termination of insulin infusion at nadir to reach plasma glucose level 4.0 mmol/L | After 12 weeks 2 days of treatment in each treatment period (Day 87 and Day 213)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Korsatko S, Jensen L, Brunner M, Sach-Friedl S, Tarp MD, Holst AG, Heller SR, Pieber TR. Effect of once-weekly semaglutide on the counterregulatory response to hypoglycaemia in people with type 2 diabetes: A randomized, placebo-controlled, double-blind, crossover trial. Diabetes Obes Metab. 2018 Nov;20(11):2565-2573. doi: 10.1111/dom.13422. Epub 2018 Jul 16. PMID 29893488
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com